CLINICAL TRIAL: NCT06358040
Title: Use of a Novel Device to Dispense Postoperative Opioids in Patients Undergoing Microdiscectomy/Laminectomy: A Pilot Study
Brief Title: Opioid Dispenser for Microdiscectomy/Laminectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0328
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use; Pain, Postoperative; Medical Device; Laminectomy; Diskectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard Opioid Pill Bottle with App (Active Comparator)
  Interventions: Other: App; Other: Standard Opioid Pill Bottle
- Opioid-Dispensing Device with App (Experimental)
  Interventions: Device: Opioid-Dispensing Device; Other: App

INTERVENTIONS:
Device: Opioid-Dispensing Device — Addinex Opioid-Dispensing Device
  Other Names: Addinex
  Arms: Opioid-Dispensing Device with App
Other: App — Addinex App
  Other Names: Addinex
Other: Standard Opioid Pill Bottle — Standard Opioid Pill Bottle
  Arms: Standard Opioid Pill Bottle with App

SUMMARY:
The opioid crisis continues to plague the United States. While great strides have been made nationwide to decrease overprescribing, improvements are still needed to appropriately educate patients on the safe and responsible use, storage and disposal of opioids. Pain after surgery is often treated with opioid medications. Opioid medications can have side effects. Some side effects are relatively minor (constipation, nausea, vomiting), while others are more severe (sedation, abnormal breathing, etc.) and can lead to serious illness or death. Opioid pain medications when used the wrong way may also be addictive. Due to theses side effects, sometimes patients feel uncomfortable about taking these medications, and doctors prescribe them very cautiously. However, when used properly and safely, opioid pain medications are excellent pain relievers.

Addinex, a technology company, has developed a device to help patients take opioids more safely. In this study the investigators aim to enroll a total of 30 patients who undergo spine surgery. Half will be randomly assigned to receive a standard pill bottle with opioids at discharge and will download a mobile app so that they can record their daily pain scores and the number of opioids they take for two weeks after surgery. The other half will receive the new opioid dispenser filled with opioids and a mobile app that generates a passcode that opens that device only at designated times. For this group of patients, every time the patient wants to take an opioid, they need to go to the app, enter their pain score before the app generates a passcode. The investigators will be tracking all study patients' opioid use and pain scores for the two weeks after surgery, will count how many pills they have left over 14 days after their surgery during a live telehealth session, and ask patients how they liked using the device. Results from this study will help understand if the Addinex device could potentially be useful to patients in the future after surgeries as opposed to typical pill bottles.

ELIGIBILITY:
Inclusion Criteria:

* opioid-naive patients or intermittent opioid users within 3 months of scheduled surgery
* At least 18 years old
* presenting for primary elective one-level lumbar laminectomy and/or discectomy via posterior approach with participating surgeon
* planned discharge on day of surgery/23 hour admission
* planned discharge to home

Exclusion Criteria:

* patients with opioid-tolerance
* patients without a smart-phone or without the ability to perform Telehealth visits
* patients unable to utilize the medication dispensing device
* patients presenting for other surgeries/surgeries with combined anterior/lateral approaches
* patient refusal
* allergy or intolerance to opioids
* planned admission after surgery
* planned discharge disposition to nursing facility or skilled rehabilitation
* planned use of or preference for opioid other than oxycodone
* patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative Opioid Consumption at Postoperative Day 14 (POD14) | Hospital Discharge to Postoperative Day 14
  Cumulative Opioid Consumption at Postoperative Day 14 (POD14) following lumbar decompression (microdiscectomy/laminectomy), expressed as number of tablets and morphine equivalents (MED in mg) and collected via app starting at discharge to 14 days later.

SECONDARY OUTCOMES:
NRS pain intensity ratings | PACU; Daily after Hospital Discharge: Postoperative Day 1 up to Postoperative Day 14
  Numerical Rating Scale (NRS) Pain Intensity Ratings from 0-10, with 0 being no pain to 10 being the worst pain possible: patient-reported in app
Patient satisfaction with the app and with the dispensing device | Postoperative Day 14
  Satisfaction survey - Device group patients will rate statements on a 5-point scale, from 1 (strongly disagree) to 5 (strongly agree)
Frequency of reported difficulties using the device | Daily up to Postoperative Day 14
  Frequency of reported difficulties using the device assessed via initiation of patient call to study team; activation of device unlocking mechanism.
Frequency of reported difficulties using the app | Daily up to Postoperative Day 14
  Frequency of reported difficulties using the app assessed via initiation of patient call/email to study team.
Opioid prescription refill rates | 6 weeks postoperatively
  Opioid prescription refill rates using electronic health records
Concordance of app data and medication left in the device or pill bottle (medication reconciliation) | Postoperative Day 14
  At Postoperative Day 14, the number of pills consumed as documented via the app, compared to actual pills left over in the device/pill bottle (telemedicine medication reconciliation).
Generation of one-time use over-ride code | Daily up to Postoperative Day 14
  Device group: Generation of one-time use over-ride code to dispense one opioid tablet, assessed via email to study team

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kramskiy, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: For researchers who provide a methodologically sound proposal and analyses to achieve aims in the approved proposal. Proposals should be directed to siderisa@hss.edu. To gain access, data requestors will need to sign a data access agreement.